CLINICAL TRIAL: NCT05624606
Title: Safety and Immunogenicity of Quadrivalent Influenza mRNA Vaccine MRT5410 in Adults Aged 18 Years and Older
Brief Title: Safety and Immunogenicity of Quadrivalent Influenza mRNA Vaccine MRT5410 in Adult Participants 18 Years of Age and Older
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAV00020; U1111-1275-1516 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Influenza Immunization
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Sentinel Cohort: Open label
  Main Cohort:
  * Open label (Sponsor, except laboratory testing personnel)
  * Blinded (Sites, except for those preparing/administering study intervention)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a parallel-group prevention study with up to 6 arms that will be blinded to participants, investigators / sub-investigators, outcomes assessors, and laboratory personnel (with the exception of the sentinel safety portion of the study, which will be open-label). The Sponsor study staff will be unblinded (except laboratory testing personnel).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Group 1: Quadrivalent Influenza mRNA Vaccine MRT5410 low dose (Experimental): participants will receive a single dose (low) of QIV mRNA vaccine
  Interventions: Biological: Quadrivalent Influenza mRNA Vaccine MRT5410
- Group 2: Quadrivalent Influenza mRNA Vaccine MRT5410 medium dose (Experimental): participants will receive a single dose (medium) of QIV mRNA vaccine
  Interventions: Biological: Quadrivalent Influenza mRNA Vaccine MRT5410
- Group 3: Quadrivalent Influenza mRNA Vaccine MRT5410 high dose (Experimental): participants will receive a single dose (high) of QIV mRNA vaccine
  Interventions: Biological: Quadrivalent Influenza mRNA Vaccine MRT5410
- Group 4: RIV4 (Active Comparator): participants will receive a single dose of RIV4 vaccine
  Interventions: Biological: Quadrivalent Recombinant Influenza vaccine RIV4
- Group 5: QIV-SD (Active Comparator): participants will receive a single dose of QIV-SD vaccine
  Interventions: Biological: Quadrivalent Inactivated Influenza Standard Dose QIV-SD
- Group 6: QIV-HD (Active Comparator): participants will receive a single dose of QIV -HD vaccine
  Interventions: Biological: Quadrivalent Inactivated Influenza High Dose QIV-HD

INTERVENTIONS:
Biological: Quadrivalent Influenza mRNA Vaccine MRT5410 — Pharmaceutical form: Liquid frozen solution for injection in a vial Route of administration: Intramuscular
  Arms: Group 1: Quadrivalent Influenza mRNA Vaccine MRT5410 low dose; Group 2: Quadrivalent Influenza mRNA Vaccine MRT5410 medium dose; Group 3: Quadrivalent Influenza mRNA Vaccine MRT5410 high dose
Biological: Quadrivalent Recombinant Influenza vaccine RIV4 — Pharmaceutical form: Liquid suspension for injection in prefilled syringe Route of administration: Intramuscular
  Other Names: Flublok Quadrivalent®
  Arms: Group 4: RIV4
Biological: Quadrivalent Inactivated Influenza Standard Dose QIV-SD — Pharmaceutical form: Liquid suspension for injection in prefilled syringe Route of administration: Intramuscular
  Other Names: Fluzone Quadrivalent®
  Arms: Group 5: QIV-SD
Biological: Quadrivalent Inactivated Influenza High Dose QIV-HD — Pharmaceutical form: Liquid suspension for injection in prefilled syringe Route of administration: Intramuscular
  Other Names: Fluzone High-Dose Quadrivalent®
  Arms: Group 6: QIV-HD

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a single intramuscular (IM) injection of up to 3 dose levels of Quadrivalent Influenza mRNA Vaccine MRT5410 compared to an active control (QIV SD, QIV HD [adults ≥ 65 years of age only], or RIV4) in adults 18 years of age and older.

DETAILED DESCRIPTION:
Approximately 12 months

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years on the day of inclusion (US) and aged 21 years on the day of inclusion (Puerto Rico)
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile OR Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 12 weeks after study intervention administration.

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Previous history of myocarditis, pericarditis, and / or myopericarditis
* Self-reported thrombocytopenia, contraindicating IM vaccination based on Investigator's judgment
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination based on Investigator's judgment
* Moderate or severe acute illness / infection (according to Investigator's judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of vaccination. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Self-reported or documented seropositivity for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus NOTE: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with immediate adverse events (AEs) | Within 30 minutes after injection
  Unsolicited systemic AEs that occur within 30 minutes after vaccination
Number of participants with solicited injection site reactions or systemic reactions | Within 7 days after injection
  Adverse reactions pre-listed in the protocol and case report form (CRF) Injection site reactions: pain, redness, swelling, hardening, bruising Systemic reactions: fever, headache, malaise, myalgia, arthralgia, chills
Number of participants with unsolicited AEs | Within 28 days after injection
  AEs that do not fulfill the conditions of solicited reactions
Number of participants with medically attended adverse events (MAAE)s | Within 180 days after injection
  AEs with a new onset or a worsening of a condition that prompts the participant or participant to seek unplanned medical advice at a physician's office or Emergency Department
Number of participants with serious adverse events (SAEs) | From Day 1 until Day 366
  SAEs reported throughout the study
Number of participants with out-of-range biological test results | Within 8 days after injection
  Out-of-range biological test results (including shift from baseline values)
Individual Hemagglutination inhibition (HAI) titer | Day 1 and Day 29
  Antibody titers are expressed as GMTs at baseline and post-baseline
Percentage of participants with detectable antibody HAI titers greater than or equal to (≥) 10 [1/dil] | Day 1 and Day 29
Individual HAI titer ratio | Day 1 and Day 29
  Ratios of antibody titers measured by HAI in each group before and after vaccination
Number of participants archiving HAI seroconversion against Antigens | Day 1 and Day 29
  Number of participants with titer < 10 [1/dil] at Day 1 and post-vaccination titer ≥ 40 [1/dil] at Day 29, or titer ≥ 10 [1/dil] at Day 1 and a ≥ 4-fold-rise in titer [1/dil] at Day 29
Percentage of participants with antibody HAI titers greater than or equal to (≥) 40 [1/dil] | Day 29
Percentage of participants with 2-fold and 4-fold rise in HAI titers | Day 1 and Day 29

SECONDARY OUTCOMES:
Neutralizing Ab titers | Day 1 and Day 29
  Neutralizing Ab titers expressed as GMTs
Individual neutralizing antibodies titer ratio | Day 1 and Day 29
Percentage of participants with 2-fold and 4-fold increase in neutralizing titers | Day 1 and Day 29
Individual HAI Ab titer ratio | Day 1, Day 91, Day 181 and Day 366
Percentage of participants with antibody HAI titers greater than or equal to (≥) 40 [1/dil] | Day 91, Day 181 and Day 366
Individual antibodies HAI titer ratio | Day 1, Day 91, Day 181 and Day 366

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (25):
- United States (23):
  - Joint Clinical Trials Huntington Park Site Number : 8400032, Huntington Park, California
  - Long Beach Clinical Trials Site Number : 8400056, Long Beach, California
  - Velocity Clinical Research, North Hollywood Site Number : 8400063, North Hollywood, California
  - California Research Foundation Site Number : 8400001, San Diego, California
  - SIMEDHealth, LLC Site Number : 8400042, Gainesville, Florida
  - Indago Research and Health Center Site Number : 8400002, Hialeah, Florida
  - Research Centers of America Site Number : 8400011, Hollywood, Florida
  - Florida International Research Center Site Number : 8400009, Miami, Florida
  - Palm Beach Research Center Site Number : 8400041, West Palm Beach, Florida
  - Velocity Clinical Research Site Number : 8400024, Meridian, Idaho
  - Brengle Family Medicine Site Number : 8400040, Indianapolis, Indiana
  - AMR Lexington Site Number : 8400035, Lexington, Kentucky
  - Meridian Clinical Research Site Number : 8400017, Norfolk, Nebraska
  - Velocity Clinical Research Site Number : 8400034, Omaha, Nebraska
  - WR-CRCN, LLC Site Number : 8400060, Las Vegas, Nevada
  - Coastal Carolina Research Center - N Charleston Site Number : 8400007, North Charleston, South Carolina
  - AMR Knoxville Site Number : 8400021, Knoxville, Tennessee
  - Elligo Health Research, Inc. Site Number : 8400037, Austin, Texas
  - Tekton Research, Inc Site Number : 8400051, Austin, Texas
  - DM Clinical Research Site Number : 8400046, Humble, Texas
  - Clinical Trials of Texas, Inc. - PPDS Site Number : 8400043, San Antonio, Texas
  - DM Clinical Research - Sugar Land Site Number : 8400045, Sugar Land, Texas
  - Martin Diagnostic Clinic Site Number : 8400058, Tomball, Texas
- Puerto Rico (2):
  - Investigational Site Number : 6300002, Barrio Sabana
  - Investigational Site Number : 6300001, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org